CLINICAL TRIAL: NCT01443715
Title: A Stepped Care Model of Adolescent Depression Treatment in Primary Care
Acronym: SCIPT-A
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6432; 1R34MH091320-01A1 (NIH)
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2013-04

CONDITIONS: Major Depressive Disorder; Dysthymia
Keywords: MDD; Dysthymia; Depressive Disorder Not Otherwise Specified (DDNOS)
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stepped Care IPT-A - Interpersonal Psychotherapy (Experimental): IPT-A focuses on communication and problem-solving skills.
  Interventions: Behavioral: Stepped Care IPT-A (SCIPT-A)
- Treatment as Usual (Active Comparator): Treatment as Usual is the standard treatment received in the community
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Stepped Care IPT-A (SCIPT-A) — Interpersonal Psychotherapy for adolescents (IPT-A) is a guideline based treatment with established efficacy focusing on reducing depression symptoms and current interpersonal problems associated with depression.
  Arms: Stepped Care IPT-A - Interpersonal Psychotherapy
Behavioral: Treatment as Usual — Standard treatment in the community
  Arms: Treatment as Usual

SUMMARY:
It is challenging for depressed adolescents and their families to access specialized mental health services. A viable option is delivering treatment in the primary care clinic (PCC) setting; however, few effective models are currently available. The overall aim of this study is to assess in the pediatric PCC, the preliminary acceptability and feasibility of a novel collaborative stepped care model of treatment for depressed adolescents.

DETAILED DESCRIPTION:
Interpersonal Psychotherapy for adolescents (IPT-A) is a guideline based treatment with established efficacy focusing on reducing depression symptoms and current interpersonal problems associated with depression. This stepped care model (SCIPT-A) first delivers a low intensity 6 session plus two parent session adaptation of IPT-A, a treatment designed for mild to moderate adolescent depression with impairment. The second phase in the model is for adolescents with persistent depressive symptoms who will receive 8 more sessions of IPT-A in combination with the addition of an antidepressant. The social worker clinicians (SW) currently employed in the PCC will be trained to deliver the Brief Interpersonal Psychotherapy for adolescents (BIPT-A)and in the second phase, the pediatrician will provide the medication treatment in collaboration with the SW clinician continuing to provide IPT-A. Fifty adolescents identified by their primary care pediatrician and meeting criteria for DSM-IV major depression, dysthymic disorder, or depression, not otherwise specified will be randomized to receive either treatment as usual (TAU) or the SCIPT-A model of stepped collaborative depression care in the PCC for 16 weeks. TAU consists of pediatrician referral of depressed adolescents to either a psychologist, social worker or child psychiatrist within the clinic or to another mental health agency in the community. All adolescents will be administered clinical interviews and self-report questionnaires during the 16 week protocol to assess treatment acceptability, feasibility, safety and preliminary change in symptoms. The project will provide information concerning the feasibility and acceptability of this treatment model for adolescent depression delivered by pediatricians and social work clinicians in pediatric primary care practice.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 13-20 years
* English and Spanish speaking adolescent
* Parent may be monolingual or bilingual in Spanish
* DSM-IV diagnosis of Major Depressive Disorder, dysthymia, or Depressive Disorder Not Otherwise Specified
* Moderate impairment in functioning
* Moderate depression severity
* Willing to refrain from other medications unless provided by investigator or PCP during the study

Exclusion Criteria:

* Diagnoses of Post Traumatic Stress Disorder , Obsessive Compulsive Disorder, current Substance abuse, Schizophrenia, bipolar disorder, Conduct disorder, Active eating disorder, Pervasive Developmental Disorder, Autism, Asberger's, Psychosis
* Engagement in severe self-injurious behavior in past 3 months
* Active suicidal ideation with plan or intent
* Mental retardation or severe learning disability
* Medical illness that may interfere with treatment
* Open Administration for Children's Services (ACS) case
* Pregnancy
* Already receiving psychotherapy or medication treatment for depression or have begun a medication trial for another diagnosis within the previous three months
* History of intolerance to fluoxetine or escitalopram
* Failed 2 completely adequate and documented Antidepressant trials
* Co-morbid Attention Deficit Hyperactivity Disorder if not on stable dose of stimulants

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2011-09; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Feasibility based on proportionality | Up to 16 weeks
  The investigators will demonstrate the feasibility of the model by calculating the proportion of: 1) adolescent who attend SCIPT-A sessions, 2) adolescents stepped to Phase II who attend their pediatric appointments for medication management, 3) adolescents in Phase II who accepted and followed the medication treatment recommendation, 4) social workers' who were willing and able to learn the SCIPT-A model as demonstrated by displaying fidelity to the treatment model.

SECONDARY OUTCOMES:
The proportion of adolescents who agree to be randomized and enrolled in the study protocol | Up to 16 weeks
  Acceptability of randomization will be determined by the proportion of adolescents from the total eligible who agree to be randomized and enrolled in the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mufson, Ph.D., Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States